CLINICAL TRIAL: NCT00714792
Title: Pilot Study: Is Overactive Bladder Caused by Subacute Urinary Tract Infections?
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 23123
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with urge incontinence due to overactive bladder
- 2: women with no urge symptoms

SUMMARY:
The purpose of this study is to look for evidence of bacteria in the urine or bladder of people with overactive bladder. Because you do not have overactive bladder, your participation in this study will be used as a comparison to those who have overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Urge urinary incontinence based on clinical history and bladder diary; subjects must have 3 or more urge incontinence episodes/day and 10 or more voids/day.
* 21 years or older
* Healthy volunteers for control subjects

Exclusion Criteria:

* Active cystitis performed on a catheterized urine specimen
* Known or suspected correctable etiology for her urge incontinence
* History of urinary tract stones, foreign bodies or malignancy
* History of recurrent Urinary Tract Infections
* Pregnant women, children
* Evidence of urge urinary incontinence or more than 1 episode of stress incontinence/day by control subject

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urogynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Flynn, MD, Principal Investigator — University of Rochester
Locations (1):
- Urogynecology and Reconstructive Pelvic Surgery Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overactive Bladder Subjects: Subjects with urge incontinence due to overactive bladder
- Control Subjects: Control subjects
Period: Overall Study
Arm/Group | Overactive Bladder Subjects | Control Subjects
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overactive Bladder Subjects | Control Subjects | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (14.3) | 54 (12.4) | 60 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Evidence of Bacteria in Urine Sample by Microbiologic Evaluation
Description: Sterile specimens were obtained from subjects. The urethra was prepared with Betadine and an 8Fr urethral catheter passed into the bladder and urine obtained in a sterile container. Bladder washings were obtained after urine was completely emptied from the bladder via the catheter. Saline (60ccs) was used to vigorously irrigate the bladder 2-3 times through the 8 Fr catheter. The bladder washings were then collected and placed in a sterile container. The experimental cultures included 100ml inoculated on Blood Agar, MacConkey Agar and Brucella Blood Agar, incubated for 72 hours at 35-37 C in ambient atmosphere supplemented with 5-8% carbon dioxide. Colonies were counted to quantify the cfu/ml and all growth of any organism was reported. Organisms were then identified using standard microbiologic techniques.
Time Frame: within one week of enrollment
Population: One overactive bladder subject had greater than 100,000 cfu in routine culture and their specimens were excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | Overactive Bladder Subjects | Control Subjects
Number analyzed (Participants) | 9 | 8
participants | 8 | 1

ADVERSE EVENTS:
Arm/Group | Overactive Bladder Subjects | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No